CLINICAL TRIAL: NCT03043300
Title: A Pilot Study to Assess the Intestinal MicroBiota Diversification States and Changes in U.S. Travelers After Return From Short-Term Travel to an Overseas South(East) Asian Destination
Brief Title: A Pilot Study Assessing Intestinal Microbiota Diversification and Changes After Travel to South(East) Asia From the US
Acronym: ABROAD
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colleen S Kraft, MD, MSc, Associate Professor, Emory University
Other Study IDs: IRB00092426; 16IPA1609428 (Other Grant/Funding Number: Centers for Disease Control and Prevention (CDC))
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Dysbiosis
Keywords: Travelers' diarrhea; Intestinal microbiota; Antibiotic resistance; Antibiotics; Gastrointestinal disorders; Infectious diseases; International Travel; Travel Medicine; Resistome; Microbiome
MeSH Terms: conditions — Dysbiosis; Gastrointestinal Diseases; Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Every stool specimen will be collected by the participant and placed in a kit and stored for deoxyribonucleic acid (DNA) extraction and sequencing. Specimens will be batched for analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- US Travelers to South or Southeast Asia: Adult individuals who are planning a short term trip to South or Southeast Asia and meet all eligibility criteria will complete the questionnaires and/or provide stool specimens at the following time points:
  1. No greater than 4 weeks prior to travel departure: Screening Criteria Review
  2. One week prior to travel departure: Pre-Travel Questionnaire and Pre-Travel Stool Specimen Collection
  3. Two weeks after return from travel: Short-Term Post-Travel Questionnaire and Short-Term Post-Travel Stool Specimen Collection
  4. 14 weeks after return from travel: Long-Term Post-Travel Questionnaire and Long-Term Post-Travel Stool Specimen Collection
  Interventions: Other: Screening Criteria Review; Other: Pre-Travel Questionnaire; Other: Pre-Travel Stool Specimen Collection; Other: Short-Term Post-Travel Questionnaire; Other: Short-Term Post-Travel Stool Specimen Collection; Other: Long-Term Post-Travel Questionnaire; Other: Long-Term Post-Travel Stool Specimen Collection

INTERVENTIONS:
Other: Screening Criteria Review — The screening criteria review is an 8 item instrument collecting information during screening about overall health, including self-reported chronic intestinal conditions, immunocompromising conditions, the use of certain medication types (immunosuppressives and antibiotics), and pregnancy status. The instrument will also collect dates of planned travel to South(east) as well as preferred dates for study visits and reminder contacts.
  This instrument will be administered verbally by the study team and completed no more than 4 weeks prior to travel departure from the United States.
  Other Names: Appendix A
Other: Pre-Travel Questionnaire — The pre-travel questionnaire is a 29 item instrument collecting information about baseline characteristics, dietary habits, travel plans, and health history.
  This questionnaire will be administered verbally by the study team and completed 1 week prior to travel departure from the United States.
  Other Names: Appendix C
Other: Pre-Travel Stool Specimen Collection — The pre-travel stool specimen collection will occur 1 week prior to travel departure from the United States.
  The processing and analyses of this stool specimen will be performed by the Centers for Disease Control and Prevention.
Other: Short-Term Post-Travel Questionnaire — The short-term post-travel questionnaire is a 19 item instrument collecting information about dates and locations of travel, food and beverages consumed while traveling, and illnesses during or following traveling.
  This questionnaire will be administered verbally by the study team and completed 2 weeks after returning to the United States from travel.
  Other Names: Appendix D
Other: Short-Term Post-Travel Stool Specimen Collection — The short-term post-travel stool specimen collection will occur 2 weeks after returning to the United States from travel.
  The processing and analyses of this stool specimen will be performed by the Centers for Disease Control and Prevention.
Other: Long-Term Post-Travel Questionnaire — The long-term post-travel questionnaire is a 16 item instrument collecting information about illnesses since last study visit, dietary habits since last study visit, and any traveling since the last visit.
  This questionnaire will be administered verbally by the study team and completed 14 weeks after returning to the United States from travel.
  Other Names: Appendix E
Other: Long-Term Post-Travel Stool Specimen Collection — The short-term post-travel stool specimen collection will occur 14 weeks after returning to the United States from travel.
  The processing and analyses of this stool specimen will be performed by the Centers for Disease Control and Prevention.

SUMMARY:
This prospective, observational pilot study is designed to assess feasibility, refine the target population, and quickly test qualitative and quantitative changes in the microbiome after short-term travel to South or Southeast Asia, regions where rates of travelers' diarrhea and intestinal colonization with antimicrobial resistant bacteria are highest.

To measure the diversity change of the intestinal microbiota, participants will complete a questionnaire and provide a stool specimen at three different time points: prior to traveling, two weeks after returning from traveling, and 14 weeks after returning from traveling.

DETAILED DESCRIPTION:
Travelers' diarrhea is the most common illness experienced by those going overseas. Estimates vary, but incidence has been reported to range between 30-60%, depending on travel destination and season. Multiple organisms have been implicated as causes of travelers' diarrhea, but bacteria account for 80-90% of cases. There is mounting evidence that the integrity of the intestinal microbiome may be a strong modulator of diarrheal disease, and that intestinal infections and other factors, including stress, antibiotic exposure, and diet may disrupt the diversity and overall composition of the microbiome. Dysbiosis, a state of altered microbiota diversity, may be less resistant to the acquisition of intestinal pathogens and colonization of multiple drug resistant organisms. Furthermore, disruptions in the microbiome that may result from an episode of travelers' diarrhea may have a role in the development of chronic diarrhea and post-infectious irritable bowel syndrome.

This prospective, observational pilot study is intended to obtain preliminary data to support the rationale for a subsequent larger cohort study. This study is designed to assess feasibility, refine the target population, and quickly test qualitative and quantitative changes in the microbiome after short-term travel (seven to 21 days) to South or Southeast Asia, regions where rates of travelers' diarrhea and intestinal colonization with antimicrobial resistant bacteria are highest.

The target population will include 10 Emory University students and/or Emory University Hospital TravelWell Clinic (TWC) patients who have international travel plans. Consented, willing, and eligible participants will complete an initial eligibility screening, followed by pre-travel, short-term post-travel, and long-term post-travel study visits. To determine specific factors associated with diversity change of the intestinal microbiota and changes in the presence of genes that code for antibiotic resistance, questionnaires designed to collect data on demographics, medical history, diet, food intake, recent (within 12 weeks of pre-travel assessment, during travel, or post-travel) illness history, medication use, travel itinerary, travel activities, and relevant food and water risk behaviors will be completed at each study visit. A stool sample will also be provided at each time point. Participants may also choose to take part in an optional sub-study which involves banking leftover stool for future research use.

The primary protocol objective is to pilot a study investigating the association between travel and changes in the intestinal microbiome (including both bacterial and fungal components) and the bacterial and fungal resistome.

The secondary protocol objective is to assess microbiota profile changes and reversion to or toward the pre-travel state by comparing pre-travel stool specimen sequencing results to short-term post-travel and long-term post-travel stool specimen sequencing results.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document.
2. Ability and willingness to comply with study protocol requirements.
3. Completed screening criteria.
4. Departure date for international travel is planned for 4 weeks from the date of informed consent.
5. Duration of international travel is planned for a minimum of seven days and maximum of 21 days.
6. International travel is planned to at least one of the following countries of South(east) Asia:

   1. South Asia, defined as: Afghanistan, Bangladesh, Bhutan, India, Maldives, Nepal, Pakistan, Sri Lanka
   2. Southeast Asia, defined as: Cambodia, Laos, West Malaysia (excluding Malaysian Borneo), Myanmar (Burma), Thailand, Vietnam

Exclusion Criteria:

1. Women of childbearing potential who self-report to be either:

   1. Currently pregnant
   2. Planning a pregnancy during study participation
2. Current diarrhea (defined as ≥ 3 unformed loose stools in 24 hours)
3. Prior episode of diarrhea (defined as ≥ 3 unformed loose stools in 24 hours) in the 12 weeks prior to date of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Emory University students and/or Emory University Hospital's TravelWell Center patients with international travel plans
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Predominant Intestinal Microbiota Genus or Strain | Pre-travel to 14 Weeks Post-Travel
  A genus of strain will be considered predominant if it represents at least 30% of all genus or strains of microbiota within the stool sample.
Change in Alpha and Beta Diversity of Intestinal Microbiota | Pre-travel to 14 Weeks Post-Travel
  Maximum percentage of all genes identified included within the same taxon will be determined from each stool sample.
Change in Firmicutes:Bacteroides Ratio of Microbiota | Pre-travel to 14 Weeks Post-Travel
  Firmicutes and Bacteroides are groups of bacteria present in the gut and the Firmicutes to Bacteroidetes ratio is considered a significant aspect of microbiota composition. The Firmicutes to Bacteroidetes ratio will be determined from each stool sample.
Change in Enteropathogens of Stool Microbiota | Pre-travel to 14 Weeks Post-Travel
  The presence of enteropathogens in stool samples will be examined pre- and post-travel.
Change in Stool Resistome | Pre-travel to 14 Weeks Post-Travel
  Review of the resistome will include a summary of the overall number and diversity of bacterial and fungal resistance genes including any new acquisition.

SECONDARY OUTCOMES:
Reversion toward pre-travel microbiota state | Pre-travel to 14 Weeks Post-Travel
  Microbiota profile changes and reversion to or toward the pre-travel state will be assessed by comparing pre-travel stool specimen sequencing results to short-term post-travel and long-term post-travel stool specimen sequencing results.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen S Kraft, MD, MSc, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Univeristy Hospital Midtown, TravelWell Center, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No